CLINICAL TRIAL: NCT02697539
Title: "Efficacy of a New Carbonate/Hydroxyapatite Nanocrystal Dentifrice on the Dental Plaque Index and the de Novo Plaque Formation Rate in Individuals Suffering From Gingivitis and/or Periodontitis"
Brief Title: Plaque Formation Rate and Toothpaste
Acronym: PFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Ehmke, Prof. Dr., University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BR-UM-01-2011
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Meridol; gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AmF/SnF2 group (Placebo Comparator): Patients in this arm were adviced to use a standart dentifrice over the course of the study (AmF/SnF2, Meridol®, GABA, Lörrach, Germany).
  Interventions: Other: mHA
- mHA group (Active Comparator): Patients in this arm were adviced to use the new dentifrice over the course of the study (mHA, BioRepair®, Wolff, Bielefeld, Germany).
  Interventions: Other: AmF/SnF2

INTERVENTIONS:
Other: AmF/SnF2 — AmF/SnF2 dentifrice used twice daily for 2 minutes for 12 weeks
  Other Names: Meridol®, GABA, Lörrach, Germany
  Arms: mHA group
Other: mHA — microcrystalline zinc-hydroxyapatite (mHA) dentifrice dentifrice used twice daily for 2 minutes for 12 weeks.
  Other Names: BioRepair® toothpaste, Kurt Wolff GmbH, Bielefeld, Germany.
  Arms: AmF/SnF2 group

SUMMARY:
This 12-week prospective, randomized, double-blind, two-center trial evaluated the impact of a microcrystalline zinc-hydroxyapatite (mHA) dentifrice on plaque formation rate (PFR) in periodontitis patients. The investigators hypothesized that mHA precipitates cause delayed plaque development when compared to a fluoridated control (AmF/SnF2), and therefore would improve periodontal health.

DETAILED DESCRIPTION:
Study Objectives and Purpose The purpose of this study is to assess the clinical efficacy of a new dentifrice, containing carbonate/hydroxyapatite nanocrystals (BioRepair®, Kurt Wolff, Bielefeld, Germany), in subjects suffering from severe gingivitis and/or mild to moderate chronic periodontitis and receiving non-surgical periodontal therapy. Clinical efficacy will be evaluated regarding clinical and microbiological parameters and compared to the use of a zinc-fluoride containing dentifrice (Meridol®, GABA, Lörrach, Germany) serving as a positive control.

Research Questions

This three-month clinical trial is conducted to answer the following research questions:

Primary Question

1. Is there a difference in de novo plaque formation as measured by the Plaque Formation Rate Index (Axelsson 1991) between subjects using the new carbonate/hydroxylapatite nanocrystal dentifrice and those using the established zinc-fluoride containing control dentifrice? Secondary Questions
2. Are there differences between subjects using the two dentifrices with respect to their subjective perception of therapy?
3. Are there differences between the two dentifrices with respect to the following periodontal measurements: change of full mouth plaque scores (O'Leary Plaque Control Record, O'Leary 1972), gingival index (Löe 1967), change of pocket probing depths (PPD's), and the percentage of sites with attachment gain of ≥ 2 mm?
4. Are there qualitative and quantitative changes regarding the composition of the oral microflora?

Study design The investigation is designed as a double blind, parallel group, and randomized trial over a 3-months period (primary endpoint). Secondary endpoints are not scheduled. Seventy-five subjects will be enrolled in this four-visit study; visits 1-4 are required for each subject. Test and control group subjects will be treated following identical therapy protocols, except for the dentifrice. Participating study centers will be the Department of Periodontology at the University of Münster and the Department of Periodontology at the University of Würzburg.

Subject Registration and Randomization Subjects that fulfil all the inclusion criteria, do not meet any exclusion criteria, and have signed the informed consent will be registered into the study by the centers Münster or Würzburg (visit 1). At visit 2 study subjects will be randomly assigned to the test group using the carbonate/hydroxyapatite nanocrystal dentifrice or the control group using a zinc-fluoride containing dentifrice. Patient randomization is warranted by using a randomization list (block randomization with 4 subjects per block). Designation of a study subject as a smoker/non-smoker will be based on recording carbonmonoxide concentration in exhaled air (non-smoker: less than 3 ppm CO in exhaled air; smoker: equal to or more than 3 ppm).

Treatment of subjects At visit 1 ("Screening/Recruitment") all subjects are informed about the projected trial. If subjects are willing to participate, they receive periodontal screening examination (PSI) and medical history is asked. At visit 2 ("Baseline", consist of two appointments at intervals of 24 hours) within the first appointment, subjects are randomized and periodontal parameters are examined. The blinded packages of different dentifrices are dispensed to the subjects. At the end, the subjects receive routine supragingival scaling with sonic scalers and polishing with an air powder device (glycin powder). Subjects are instructed to abstain from oral hygiene for the next 24 hours. At the end, subjects fill out the two questionnaires. At the second appointment, plaque formation rate is examined and subjects are instructed to brush with their already used toothbrush for 2 minutes at least twice per day at home.

Four weeks after "Baseline" at visit 3 ("Treatment", consist of two appointments at intervals of 24 hours), periodontal parameters are examined and all subjects receive full mouth supra- and subgingival debridement in two sessions on two consecutive days. Debridement is performed with sonic scalers using micro tips under local anesthesia and polishing is performed with an air powder device. Subjects are instructed to abstain from oral hygiene for the next 24 hours. At the second appointment, plaque formation rate is examined, all subjects receive full mouth supra- and subgingival debridement, and are instructed to brush with their already used toothbrush for 2 minutes at least twice per day at home. Two months after "Treatment" at visit 4 ("Reevaluation", consist of two appointments at intervals of 24 hours) periodontal parameters are examined and all subjects receive full mouth supragingival debridement in one session. Subjects are instructed to abstain from oral hygiene for the next 24 hours. At the second appointment, plaque formation rate is examined, all subjects receive full mouth supragingival debridement. Subjects return the dentifrice packages.

Over the course of the study no medication except the dentifrice or local anesthesia is administered. During the trial, subjects are not permitted to undergo advanced periodontal treatment (i.e. periodontal surgery) or to receive drugs influencing periodontal health.

Clinical Examinations After assessing the plaque and the gingival index (O'Leary 1972, Löe 1967) clinical measurements of full mouth pocket probing depths (PPD), bleeding on probing (BOP), gingival recessions (GR), and furcation involvement are taken. All measurements, except for furcation involvement, are taken at six sites per tooth (mesiobuccal, mid-buccal, distobuccal, mesiolingual, mid-lingual and distolingual). Measurements of PPD, BOP, and GR are performed using a standard Florida Probe® handpiece (Florida Probe Corp., Gainsville, FL, USA). Clinical measurements are taken at baseline, after 4 weeks, and after 3 months (visits 2a, 3a, and 4a). Smoking habits are determined by an objective chairside measurement of carbon monoxide concentration in exhaled air (Bedfont-Smokerlyzer®, Bedfont, UK) at visits 1 through 4. Intraoral radiographs and photographs are taken at baseline.

Specification of Psychological Assessments At visits 2a and 4a patients are asked to complete the Oral Health Impact Profile - German Version (OHIP-G 49) and the German version of the Client Satisfaction Questionnaire (ZUF-8) as a standardized instrument used to measure health outcome.

Oral Health Impact Profile - German Version (OHIP-G 49) The original English version of the questionnaire was developed by Slade and Spencer (1994). The German translation and validation of the instrument was performed by John et al. (2002). The OHIP-G 49 contains 49 items that address specific problems of oral health, e.g., "problems with chewing of food" or "pain in the gums". Each item is assessed on a five-point scale (0: never to 4: very often). A sum score of all of the items is calculated as an indicator for current oral health. The completion of the questionnaire takes about ten minutes.

ZUF-8 The patients´ satisfaction with the treatment is evaluated by means of the Fragebogen zur Patientenzufriedenheit (ZUF-8, Schmidt et al. 1989) which represents the German version of the Client Satisfaction Questionnaire (CQS, Attkisson & Zwick 1982).

Microbiological Examination For microbiological analysis, pooled subgingival plaque samples are taken from four different teeth with at least one site with PPDs of ≥ 4 mm from each study subject. The pooled subgingival plaque sample is collected in a transport tube containing 500 µl Ringer-Glycerin-Solution. The pooled samples are at once taken to the laboratory for analysis or stored in liquid nitrogen.

Supragingival plaque is collected from four sites per sample tooth. From the buccal and lingual sites samples are taken using Periotron© adapted to the tooth surface to collect dental plaque from the area near the gingival margin. Interproximal, supragingival plaque samples are collected by inserting a sterile paperpoint horizontally in buccal to lingual direction near the gingival margin. Samples from buccal/lingual and from interproximal sites are pooled respectively (two pooled samples from each subject per visit 2a, 3a, 4a) in a seperate transport tube containing 500 µl Ringer-Glycerin-Solution. The pooled samples are at once taken to the laboratory for analysis or stored in liquid nitrogen.

Sample teeth are randomly selected at baseline as shown in Fig. 2 to assure equal distribution throughout the mouth, and remain the same over the course of the study. The whole bacterial counts are quantified by culture at study visits 2a, 3a, and 4a.

Laboratory Processing, Microbiological Analysis After subgingival plaque sampling, the samples are taken immediately in the laboratory for further processing or stored in liquid nitrogen until the study is finished. After finishing the trial they will be carried to Münster. For transport they are stored in carbon dioxide snow and are stored in liquid nitrogen in the laboratory in Münster again. The pooled samples are sonicated for 10 seconds (Sonotex RK 82, Bandelin Electronic AG, Berlin, Germany) and diluted in tenfold steps. 0.1 ml of the undiluted suspension and 0.1 ml aliquots of the dilutions are spread on different culture media. In parallel supragingival plaque samples are spread on CDC agar and are stored in an aerobe atmosphere at 37 degree above zero overnight.

For quantitative enumeration the undiluted and diluted suspensions are spread on non-selective blood agar (CDC agar) plates containing 5% defibrinated sheep blood supplemented with 5mg/l hemin (Merck, Darmstadt, Germany), 1 mg/l vitamin K1, and 10 mg/l N-acetylmuramine acid (NAM). NAM is supplemented for cultivation of T. forsythensis. The plates are incubated in an atmosphere containing N2 (85%), H2 (10%), and CO2 (5%) for 7 days. Total cultivable counts are assessed for each of the plaque samples. The evaluation of pooled plaque samples on CDC agar and the total cultivable counts are reported quantitatively as colony forming units (CFU/ml). In further investigation the present of specific periodontal pathogens will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pocket probing depths (PPDs) of ≥ 4 mm at a minimum of four teeth (except third molars)
* age ≤ 18 to ≤ 75 years
* at least 10 natural teeth in situ (except third molars)
* non-smokers

Exclusion Criteria:

* known systemic diseases that may influence the periodontal conditions
* regular consumption of drugs that may interfere with periodontal conditions
* undergoing or requiring extensive dental or orthodontic treatment
* pregnancy or breastfeeding
* professional periodontal therapy during 6 months prior to baseline.
* periodontal pockets ≥ 6 mm in more than 2 sextants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome plaque formation rate (PFR) was measured 24 hours after all teeth were treated mechanically. | Measured 24 hours after all teeth were treated mechanically .
  For the recording of PFR,all teeth were stained with a plaque revealer (Mira 2-Ton® Miradent, Hager & Werken GmbH, Duisburg, Germany).

SECONDARY OUTCOMES:
full mouth plaque control record (PCR, O'Leary 1972). | at baseline (visit 2a), after 4 weeks and after 12 weeks
  For the recording of PCR,all teeth were stained with a plaque revealer (Mira 2-Ton® Miradent, Hager & Werken GmbH, Duisburg, Germany). The % of sites showing bacterial plaque was measured
gingival index (GI, Löe 1967), | at baseline (visit 2a), after 4 weeks and after 12 weeks
  Inflammation grade of the ginigiva is measured. Gradual index (0-3)
pocket probing depths (PPD) | at baseline (visit 2a), after 4 weeks and after 12 weeks
  a measurement (mm) from the gingival margin to the clinical bottom of the periodontal pocket. Describes the severity of periodontal disease.
bleeding on probing (BOP, Lang et al. 1990), | at baseline (visit 2a), after 4 weeks and after 12 weeks
  If the gingiva starts to bleed after gentle probing, this is a sign of inflammation. Schould disapear after sufficient therapy. The % of sites showing bleeding is measured.
gingival recession (GR) | at baseline (visit 2a), after 4 weeks and after 12 weeks
  Measurement from the enamel-cementum-border to the gingival margin (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Ehmke, Prof. Dr., Principal Investigator — University of Münster, Department of Periodontology Waldeyerstr. 30, 48149 Münster; Ulrich Schlagenhauf, Prof. Dr., Study Director — University of Würzburg, Department of Periodontology Pleicherwall 2, 97070 Würzburg

IPD SHARING:
Plan to Share IPD: Undecided
we would provide data for meta analysies. But because this was not scheduled while prototcol approvement, this must be finally decided by the responisble ethic comittee.

REFERENCES:
- [Derived] Harks I, Jockel-Schneider Y, Schlagenhauf U, May TW, Gravemeier M, Prior K, Petersilka G, Ehmke B. Impact of the Daily Use of a Microcrystal Hydroxyapatite Dentifrice on De Novo Plaque Formation and Clinical/Microbiological Parameters of Periodontal Health. A Randomized Trial. PLoS One. 2016 Jul 28;11(7):e0160142. doi: 10.1371/journal.pone.0160142. eCollection 2016. PMID 27467683